CLINICAL TRIAL: NCT04520854
Title: Physical Rehabilitation Through Telehealth for an Ankle Sprain: A Randomized Controlled Trial
Brief Title: Telehealth Delivered Physical Rehabilitation for an Ankle Sprain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyle Kosik (Other)
Responsible Party: Sponsor-Investigator, Kyle Kosik, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 60997; #1920GGP02 (Other Grant/Funding Number: National Athletic Trainers' Association Research and Education Foundation)
Record Dates: First submitted 2020-08-12; First posted 2020-08-20 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Ankle Sprains; Telerehabilitation; Analgesic, Opioid; Analgesics, Non-narcotic; Anti-Inflammatory Agents, Non-Steroidal; Implementation Science; Acute Pain; Quality of Life
MeSH Terms: conditions — Ankle Injuries; Acute Pain

STUDY DESIGN:
Intervention Model Description: The Specific Aims will be addressed using a single-blind, parallel-am randomized control trial. The independent variables will be group (Telehealth, usual care) and time (baseline, post-intervention, 1-month follow-up). Participants assigned to the Telehealth group will complete a 2-week intervention consisting of 5 live-video sessions. A 2-week intervention will be used to allow for the normal recovery of acute symptoms and account for the average number of supervised physical rehabilitation visits (5 sessions) currently recommended. The usual care group will be instructed to follow their physicians' orders during the two-week intervention period. The dependent variables for will be assessed on the injured limb only for both groups. A Co-I will collect all dependent variables and will be blinded to group assignment.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2-week Telehealth Protocol (Experimental): Participants randomized to this arm will receive 5 live-video sessions. The first 2 live-video sessions will occur during the first week, last 20 minutes each and separated by 48-72 hours. The last 3 live-video sessions will occur during the second week, last 30-minutes each and separated by 24-48 hours.
  Interventions: Other: Telehealth Protocol
- 2-week Usual Care (Active Comparator): The usual care group will be used to reflect the current care provided to patients after discharged from the emergency department for an ankle sprain.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Telehealth Protocol — The first live-video session will orient participants to the features of the software, discuss the checklist to minimize environmental distractions, gauge how participants are managing their symptoms (pain, swelling) and provide non-pharmacological alternatives to supplement their current treatment strategies.
  The second live-video session will be used re-examine how the participant is managing their symptoms (pain, swelling) and re-emphasize non-pharmacological alternatives.
  The remaining live-video sessions will be focused on giving participants home-based therapeutic exercises. The therapeutic exercises will target the four main areas important to ankle sprain recovery: 1) range of motion; 2) balance; 3) gait; and 4) strength. All of the therapeutic exercises are based on previously published criteria for the rehabilitation of an LAS. The progression will start with single-plane, non-weight bearing or low-force activities and will advance at the same rate.
  Arms: 2-week Telehealth Protocol
Other: Usual Care — The usual care group will be instructed to follow their treating physicians' orders. Participants will not receive instructions on how to self-manage symptoms nor a home-based exercise program.
  Arms: 2-week Usual Care

SUMMARY:
A vast majority (75-85%) of ankle sprain patients treated in emergency departments (ED) receive pain medication and are not referred for physical rehabilitation. Therefore, purpose of this study is to increase access to the standard of care for an ankle sprain by provide patients with physical rehabilitation delivered through telehealth. The purpose of this study includes compare a 2-week telehealth intervention to the usual care for treating 1) subjective function; 2) physical impairments; 3) medication consumption; and 4) patient-perceived barriers. The central hypothesis is participants receiving the 2-week telehealth intervention will 1) have less pain and disability; 2) improve balance and ankle range of motion; 3) consume less medication; and 4) reports positive feedback compared to the usual care group.

DETAILED DESCRIPTION:
Musculoskeletal injuries account for 15% of all emergency department (ED) visits in the United States. More than 1 million people are treated in the ED every year for an ankle sprain; making it the most common musculoskeletal injury. Most ankle sprain patients do not receive the recommended care because the vast majority (75-85%) are prescribed opioid or non-opioid medication and are not referred for follow-up health care services. Physical rehabilitation is the gold standard for follow-up care because of its known benefits as a non- pharmacological alternative to pain management and for restoring normal function. However, ankle sprain patients aren't referred to physical rehabilitation because of the lack of access to timely health care services, particularly for rural communities or underserved urban areas. A lack of access and/or increased wait time from referral to the first outpatient visit has been associated with detrimental physical and psychological effects. In fact, without physical therapy, ankle sprain patients can develop chronic pain, become less physically active, report having a worse health-related quality of life, suffer a recurrent injury and show early symptoms of post- traumatic osteoarthritis. Telehealth is a novel method of care delivery designed to bridge this gap by leveraging live-video communication platforms to provide timely health care services. Therefore, the rationale for this project is demonstrating the benefits of telehealth to deliver the standard of care for an ankle sprain will lead to new methods providing timely access to follow-up health care services for patients discharged from the ED for not only an ankle sprain, but a wide variety of musculoskeletal injuries. The specific aims for the proposed research include comparing a 2-week telehealth intervention to the usual care for 1) treating pain, disability, health-related quality of life, and physical activity; 2) ankle range of motion, static and dynamic balance; 3) opioid and non-opioid medication consumption; and 4) the feasibility, acceptability and appropriateness of each intervention. The investigators hypothesize, compared to the usual care, participants receiving telehealth will 1) have less pain and disability; 2) a better health-related quality; 3) increased physical activity levels; 4) greater ankle range of motion; 5) better static and dynamic balance; 5) take fewer opioid and non-opioid medication; and 5) report positive feedback. A single-blind, randomized control trial will assign 70 ankle sprain patients discharged from the ED to two equal groups (Telehealth, usual-care). The telehealth intervention includes 5-live video sessions with an investigator providing education about injury management, long-term health and therapeutic exercises. The usual care group will follow their physicians' orders. The expected outcomes will illustrate the value of immediate access to rehabilitative services delivered via telehealth for an ankle sprain.

ELIGIBILITY:
Inclusion Criteria:

* All race and ethnic groups
* Men and women between 15-35 years of age
* Discharged from an ED within 72 hours of being diagnosed with a grade 1 or 2 acute lateral ankle sprain (LAS) and not receiving a physical therapy referral from their treating physician will be enrolled. A LAS will be defined as an incident in which the rearfoot was inverted and resulted in a combination of pain, swelling and time lost from activity for at least one day.
* Participants with or without a prior history of an ankle sprain will be included unless the most recent injury occurred within six months prior to enrollment. Participants with a prior history of ankle sprain will only be included if the most recent injury occurred beyond six months prior to enrollment: 1) to ensure they recovered and returned to their normal activity; 2) to ensure they are experiencing acute rather than chronic symptoms; 3) to ensure they are all exposed to similar treatment options.All race and ethnic groups will be included.

Exclusion Criteria:

* Diagnosed with a concomitant injury (e.g., fracture)
* History of lower extremity surgery, or conditions other than an ankle sprain that affect balance and gait
* Do not speak English.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale | Change from baseline at 24-72 hours immediately post intervention AND change from immediately post intervention at 1 month.
  Self-reported levels of acute ankle pain at rest, while walking, climbing stairs and when running will be recorded using separate 100 mm VAS for each of those tasks. Each VAS will be anchored on the left (0 mm) with 'no pain' and 'worst pain' on the right (100 mm). Participants will place a single handwritten mark at one point along the 100 mm line. The linear distance from the left end of the line to the participants' mark will be measured using a standard ruler and recorded in millimeters. Therefore, a higher numerical value reflects greater levels of pain intensity during the selected activity. Excellent test-retest reliability has been reported for assessing acute pain using a VAS (ICC=0.97).
Change in Foot and Ankle Ability Measure (FAAM) | Change from baseline at 24-72 hours immediately post intervention AND change from immediately post intervention at 1 month.
  The FAAM is a region-specific patient-reported outcome to measure self-reported function in patients with ankle pathologies. The FAAM contains items that measure the level of difficulty patients have performing activities of daily living (ADL) and physical activity (Sport). Items are scored on a 5-point Likert scale with 4 representing 'no difficulty' and 0 indicating 'unable to do'. The sum from both subscales is calculated and presented as a percentage of the total possible points. A lower score is indicative of decreased function and HRQL. The FAAM is reliable (ADL: ICC=0.89; Sport: ICC=0.087), valid and responsive to change after intervention.
Documentation of opioid and non-opioid medication consumed: | Total amount consumed between baseline to 24-72 hours immediately post intervention AND total amount consumed between immediately post intervention to 1 month folllow-up.
  Participants ≥18 years of age and legal guardians of adolescents will be given a daily log to record the type and dose of any opioid or non-opioid medication consumed. Frequent reminders to complete the daily medication log will be sent via email to both groups and the daily log will be collected at the end of each week. Secondly, all participants or legal guardian's will be interviewed weekly over the phone with and asked if they had filled their opioid prescription, the quantity of any medication consumed, and any new opioid prescriptions filled.
  Information gathered will be used to calculate the morphine milligram equivalent (MME) per day for any opioid medication. The MME per day consumed from baseline to post- intervention and post-intervention to the 1-month follow-up will be summed and used for statistical analysis. The number of tablets consumed per day for all non-opioid medication will be recorded, summed and used for statistical analysis.
Change in Feasibility of Intervention Measure (FIM): | Change from 24-72 hours immediately post intervention at 1 month follow-up.
  Feasibility is the extent to which a new treatment can be successfully used or implemented within a setting. The FIM contains four, 5-point Likert scales that assess the perceived feasibility of the intervention. Each Likert Scale is anchored with a 1 representing 'completely disagree' and 5 indicating 'completely agree'. The average score is calculated, with a higher score suggesting the intervention is perceived as being more feasible. The FIM has demonstrated acceptable internal consistency with a Cronbach α score of 0.89 and good test-retest reliability (r=0.88).
Acceptability of Intervention Measure (AIM) | Post-intervention and 1-month follow-up
  Acceptability is the extent to which stakeholders perceive a treatment to be palatable or satisfactory. The AIM includes four, 5-point Likert scales that assess the perceived acceptability of the intervention. Each Likert Scale is anchored with a 1 representing 'completely disagree' and 5 indicating 'completely agree'. The average score is calculated, with a higher score suggesting the intervention is perceived as being more acceptable. The AIM has shown acceptable internal consistency with a Cronbach α score of 0.85 and good test-retest reliability (r=0.80).
Intervention Appropriateness Measure (IAM) | Change from 24-72 hours immediately post intervention at 1 month follow-up.
  Appropriateness is the perceived fit, relevance and compatibility of the intervention to address a particular issue. The IAM includes four, 5- point Likert scales that assess the perceived appropriateness of the intervention. Each Likert Scale is anchored with a 1 representing 'completely disagree' and 5 indicating 'completely agree'. The average score is calculated, with a higher score suggesting the intervention is perceived as more appropriate. IAM has exhibited acceptable internal consistency with a Cronbach α score of 0.91 and good test-retest reliability (r=0.73).
Disablement in the Physical Active Scale (DPA). | Change from baseline at 24-72 hours immediately post intervention AND change from immediately post intervention at 1 month.
  The DPA is a 16-item global outcome instrument. Responses to each item are based on a 5-point Likert scale ranging from 'no problem' to 'severe'. (26) High test-retest reliability (ICC = 0.943) and internal consistent (alpha = 0.890-0.908) have been reported.
International Physical Activity Questionnaire (IPAQ)- Short Form | Change from baseline at 24-72 hours immediately post intervention AND change from immediately post intervention at 1 month.
  The IPAQ is regularly administered to quantify the kinds of physical activity that people do as part of their everyday lives. The IPAQ has been shown to be a reliable and valid measure of physical activity among all age categories.
Weight-bearing lunge test (WBLT) | Change from baseline at 24-72 hours immediately post intervention AND change from immediately post intervention at 1 month.
  Closed-kinetic chain dorsiflexion will be assessed bilaterally. A standard metric tape measure will be secured to the floor and perpendicular to a wall. Participants will stand facing the wall, with their hands on the wall and their feet in a tandem stance over the secured tape measure. Keeping their second toe and center of their heel on the tape measure, participants will be instructed to perform a forward lunge in which the anterior surface of the knee of the involved limb touches the wall. Participants will gradually be moved further away from the wall in 1 cm increments until the participant can no longer touch the wall with their anterior knee and keeping their heel on the ground. The maximum distance from the wall while continuing to maintain contact with the wall and heel on the ground will be recorded as maximum dorsiflexion ROM in cm. Three trials will be performed for each limb. \The average of the three trials for each limb will be used for statistical analysis.
Star-Excursion Balance Test (SEBT) | Change from baseline at 24-72 hours immediately post intervention AND change from immediately post intervention at 1 month.
  Dynamic balance will be assessed bilaterally. The anterior, posteromedial, and posterolateral reach directions of the SEBT will be used. Participants will maintain a single-leg stance on the involved limb while reaching for maximum distance with the non-stance limb. During the anterior reach the participant's first toe is placed at the 0 point of the tape measure, while the heel is placed at 0 on the tape measure for the posterolateral and posteromedial directions. The participant is instructed to gently touch the tape measure with the most distal part of the reaching limb while maintaining a single-leg base of support on the test limb, and then return to double-leg stance. The participant's hands must remain on their hips and the stance heel must remain in contact with the ground. Four practice trials will be performed in each direction, followed by three test trials in each direction. The average across all three trials for each direction will be used for statistical analysis.
Static Postural Control | Change from baseline at 24-72 hours immediately post intervention AND change from immediately post intervention at 1 month.
  Static balance will be assessed bilaterally. A single-limb with eyes-open balance task will be utilized. A force platform (AccuSway Plus, AMTI, Watertown, MA) integrated with Balance Clinic software (AMTI, Watertown, MA) will be used to record center of pressure (COP) trajectories in the anteroposterior (AP) and mediolateral (ML) directions at a sampling rate of 100Hz. Participants will be asked to balance in a barefoot single-limb stance on the middle of the force platform, keep their hands on the chest, and stare at an "X" in front of them while keeping their foot flat on the force plate. Participants will be allowed three practice trials and then asked to perform three testing trials with their eyes-open. Participants will be instructed to balance quietly in a single-limb stance for 20 seconds while COP data will be collected. The COP velocity (COPV) (cm/s) and measures of time-to-boundary (TTB) (sec) in each direction will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Kosik, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No